CLINICAL TRIAL: NCT00416312
Title: Dose-Response in Radioimmunotherapy of Lymphoma
Brief Title: Iodine I 131 Tositumomab or Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J0636; CDR0000522705 (Registry Identifier: PDQ (Physician Data Query)); R01CA116477-01A1 (NIH); NA_00001712 (Other: JHM IRB)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
Keywords: extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; Waldenström macroglobulinemia; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; primary central nervous system non-Hodgkin lymphoma; adult nasal type extranodal NK/T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Conventional & Patient-Specific Dosimetry: Tumor absorbed dose calculations determined using both conventional dosimetry and 3D-RD patient-specific dosimetry software.
  Interventions: Device: Patient-specific dosimetry; Device: conventional dosimetry

INTERVENTIONS:
Device: Patient-specific dosimetry — Tumor absorbed dose calculation using patient-specific 3D-RD dosimetry software.
  Patients receive dosimetric tositumomab IV over 60 minutes followed by iodine I 131 (^131I) tositumomab IV over 20 minutes on day 0. Patients undergo PET/CT scans and SPECT/CT scans on days 0; 2, 3 or 4; and 6 or 7. Patients who have acceptable biodistribution receive therapeutic tositumomab IV over 60 minutes followed by ^131I tositumomab IV over 20 minutes on approximately day 7.
Device: conventional dosimetry — Doses calculated using conventional dosimetry software.
  Patients receive dosimetric rituximab IV followed by indium In 111 (^111In) ibritumomab tiuxetan IV over 10 minutes on day 1. Patients undergo positron emission tomography (PET)/CT scans and single-photon emission computed tomography (SPECT)/CT scans between 2-24, 48-72, and 90-120 hours after ^111In ibritumomab tiuxetan administration. Patients who have acceptable biodistribution receive therapeutic rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes between days 7-9.

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies, such as iodine I 131 tositumomab and yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. This may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: This clinical trial is studying the side effects, best dose, and how well iodine I 131 tositumomab or yttrium Y 90 ibritumomab tiuxetan works in treating patients with non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the relationship between estimated absorbed dose and tumor response using different dosimetric methodologies in patients with non-Hodgkin's lymphoma treated with iodine I 131 tositumomab or yttrium Y 90 ibritumomab tiuxetan.
* Determine the relationship between estimated absorbed dose and normal organ toxicity using different dosimetric methodologies in these patients.

Secondary

* Assess the difference in the dose-response relationship between dosimetric methodologies in these patients.
* Assess the influence of prior therapy on the dose-response relationship for hematologic toxicity in these patients.

OUTLINE: Patients are stratified according to planned radioimmunotherapy treatment (iodine I 131 tositumomab vs yttrium Y 90 ibritumomab tiuxetan).

* Stratum 1: Patients receive dosimetric rituximab IV followed by indium In 111 (^111In) ibritumomab tiuxetan IV over 10 minutes on day 1. Patients undergo positron emission tomography (PET)/CT scans and single-photon emission computed tomography (SPECT)/CT scans between 2-24, 48-72, and 90-120 hours after ^111In ibritumomab tiuxetan administration. Patients who have acceptable biodistribution receive therapeutic rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes between days 7-9.
* Stratum 2: Patients receive dosimetric tositumomab IV over 60 minutes followed by iodine I 131 (^131I) tositumomab IV over 20 minutes on day 0. Patients undergo PET/CT scans and SPECT/CT scans on days 0; 2, 3 or 4; and 6 or 7. Patients who have acceptable biodistribution receive therapeutic tositumomab IV over 60 minutes followed by ^131I tositumomab IV over 20 minutes on approximately day 7.

In both strata, blood is collected at baseline to measure FLT-3 levels. All patients also undergo a baseline PET/CT scan.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 88 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-Hodgkin's lymphoma
* Measurable disease by CT scan or nuclear medicine imaging
* Eligible, by standard of care criteria, for iodine I 131 tositumomab or yttrium Y 90 ibritumomab tiuxetan treatment

PATIENT CHARACTERISTICS:

* No other malignancy within the past 3 years except basal cell carcinoma or squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No alcoholism or drug abuse within the past 2 years
* No severe emotional, behavioral, or psychiatric problems that would limit study compliance

PRIOR CONCURRENT THERAPY:

* No concurrent participation in another investigational drug study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for NHL by rituximab or zevalin
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2006-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Sgouros, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All NHL patients treated by either Bexxar or Zevalin
Period: Overall Study
Arm/Group | Conventional & Patient-specific Dosimetry
Started | 9
Conventional Dosimetry | 9
Patient-specific Dosimetry | 9
Completed | 7
Not Completed | 2
Not completed — tumors not visible on imaging | 2

BASELINE CHARACTERISTICS:
Population: Patients being treated for lymphoma using I-131-labeled antibody were imaged and tumor dosimetry was performed using conventional and patient-specific dosimetry. Tumors could not be detected on imaging for 2 of the 9 enrolled patients.
Arm/Group | Conventional & Patient-specific Dosimetry
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants] — Population: Tumors could not be detected on imaging for 2 of the 9 enrolled patients
  Participants
    number analyzed (Participants) | 7
    <=18 years | 0
    Between 18 and 65 years | 1
    >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Tumors could not be detected on imaging for 2 of the 9 enrolled patients
  Participants
    number analyzed (Participants) | 7
    Female | 1
    Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Tumor Absorbed Dose
Description: tumor absorbed dose (Gy)
Time Frame: up to 4 years
Measure: Mean (Standard Deviation); unit: Gy
Units Other Than Participants: tumor
Arm/Group | Conventional & Patient-specific Dosimetry
Number analyzed (Participants) | 7
Number analyzed (tumor) | 7
Gy
  Conventional dosimetry | 3.01 (3.04)
  Patient-specific dosimetry | 3.41 (3.1)

ADVERSE EVENTS:
Description: Adverse event data was not collected since this was a data collection study tacked on to routine patient treatment
Arm/Group | Conventional & Patient-specific Dosimetry
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No